CLINICAL TRIAL: NCT04038385
Title: WIC-Based Intervention to Promote Healthy Eating Among Low-Income Mothers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: William Paterson University of New Jersey (Other)
Responsible Party: Principal Investigator, Jennifer Di Noia, Professor, Department of Sociology, William Paterson University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1R21CA230476-01 (NIH)
Record Dates: First submitted 2019-07-14; First posted 2019-07-30 (Actual); Results first posted 2021-12-23 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-11

CONDITIONS: Cancer Prevention; Diet Modification; Vegetable Intake

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): This group will receive routine services provided by WIC and an intervention that will combine behaviorally-focused nutrition education with 1) the establishment of a WIC-based farmers' market (implemented in 2019 during the WIC Farmers' Market Nutrition Program voucher issuance period [June 19 to August 19]), and 2) monthly trips to an area farmers' market (between September 1, 2019 and November 30, 2019 [the end of the local growing season]).
  Interventions: Behavioral: Multilevel Behavioral Intervention
- Control (No Intervention): This group will receive routine services provided by WIC only.

INTERVENTIONS:
Behavioral: Multilevel Behavioral Intervention — Behaviorally-focused intervention grounded in the Social Ecological Model and Social Cognitive Theory to promote vegetable intake and the redemption of seasonal Farmers' Market Nutrition Program vouchers and monthly Cash Value Vouchers at farmers' markets.
  Arms: Intervention

SUMMARY:
Whole grains, non-starchy vegetables, fruit, and beans are a consistent feature of diets associated with a lower risk of cancer and other diet-related diseases. For cancer risk reduction, the American Cancer Society recommendation is to consume at least 2.5 cups of a variety of fruits and vegetables daily. Other than dietary choices, weight control and physical activity levels are important modifiable determinants of cancer risk. This study finalized a novel, theory-driven farm-to-WIC intervention developed in preliminary work to promote vegetable intake among low-income adults served by the Special Supplemental Nutrition Program for Women, Infants, and Children (WIC). In New Jersey (the location of the study), WIC provides participants up to $30 in seasonal Farmers' Market Nutrition Program (FMNP) vouchers and monthly cash value vouchers or CVV (valued at $11 for adults and $8 for children at the time of the study) redeemable at farmers' markets. The program combined behaviorally focused nutrition education with the establishment of a WIC-based farmers' market (implemented in the summer of 2019 during the FMNP voucher issuance period). Content to address other modifiable determinants of cancer risk was added. To create additional opportunities for experiential and hands-on learning, monthly trips to an area farmers' market were held (between September 1, 2019 [after the WIC-based market was discontinued] and November 30, 2019 [the end of the local growing season]). The research employed an experimental design to initially test the intervention in 3 WIC agency sites (1 intervention and 2 control sites) with 297 urban, primarily Hispanic adults. Program effects on primary outcomes of vegetable intake (measured objectively using dermal carotenoids as a biomarker of intake and via self-report) and FMNP voucher redemption (objectively assessed using data provided by WIC) were examined at mid- and post-intervention (3 and 6 months post-baseline, respectively). Intervention effects on potential hypothesized mediators and the redemption of CVV at farmers' markets, participant satisfaction with the program, and the cost-effectiveness of the intervention also were examined.

ELIGIBILITY:
Inclusion Criteria:

* English- or Spanish-speaking
* Farmers' Market Nutrition Program (FMNP) voucher recipient or caregiver of a child FMNP voucher recipient
* Not less than 3 months from expected delivery date (pregnant women)
* Eligible to receive WIC benefits for 6 months after study entry

Exclusion Criteria:

● Restrictions of food intake (has food allergies or foods that cannot be eaten)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 297 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2021-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Di Noia, PhD, Principal Investigator — William Paterson University
Locations (1):
- Saint Joseph's WIC Program, Paterson, New Jersey, United States

REFERENCES:
- [Background] Di Noia J, Gellermann W. Use of the Spectroscopy-Based Veggie Meter(R) to Objectively Assess Fruit and Vegetable Intake in Low-Income Adults. Nutrients. 2021 Jun 30;13(7):2270. doi: 10.3390/nu13072270. PMID 34209048
- [Result] Di Noia J, Monica D, Jensen HH, Sikorskii A. Economic evaluation of a farm-to-Special Supplemental Nutrition Programme for Women, Infants and Children intervention promoting vegetable consumption. Public Health Nutr. 2021 Aug;24(12):3922-3928. doi: 10.1017/S1368980021001981. Epub 2021 May 11. PMID 33972002
- [Result] Di Noia J, Monica D, Sikorskii A, Nelson J. Pilot Study of a Farm-to-Special Supplemental Nutrition Program for Women, Infants, and Children (WIC) Intervention Promoting Vegetable Consumption. J Acad Nutr Diet. 2021 Oct;121(10):2035-2045. doi: 10.1016/j.jand.2020.12.020. Epub 2021 Jan 22. PMID 33487590
- [Result] Di Noia J, Monica D, Sikorskii A. Process Evaluation of a Farm-to-WIC Intervention. J Acad Nutr Diet. 2021 Oct;121(10):2021-2034. doi: 10.1016/j.jand.2021.05.014. Epub 2021 Jun 16. PMID 34144918

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred from June 3, 2019, to August 1, 2019. Participants were recruited via telephone (prior to forthcoming appointments with WIC) and in person at collaborating WIC agency sites.
Groups:
- Intervention: This group will receive routine services provided by WIC and an intervention that will combine behaviorally-focused nutrition education with 1) the establishment of a WIC-based farmers' market (implemented in 2019 during the WIC Farmers' Market Nutrition Program voucher issuance period [June 19 to August 19]), and 2) monthly trips to an area farmers' market and local supermarket (between September 1, 2019 and November 30, 2019 [the end of the local growing season]).
  Multilevel Behavioral Intervention: Behaviorally-focused intervention grounded in the Social Ecological Model and Social Cognitive Theory to promote vegetable intake and the redemption of seasonal Farmers' Market Nutrition Program vouchers and monthly Cash Value Vouchers provided to WIC participants to purchase fruits and vegetables.
Period: Overall Study
Arm/Group | Intervention | Control
Started | 160 | 137
Completed (143 (intervention) and 130 (control) provided self-report data; 137 (intervention) and 124 (control) provided biometric data. For biometric data,13 (intervention) and 10 (control) competed the baseline assessment only.) | 143 | 130
Not Completed | 17 | 7
Not completed — Completed baseline assessment only | 7 | 4
Not completed — Moved out of area | 4 | 2
Not completed — Discontinued study involvement | 6 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 160 | 137 | 297
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.5 (7.2) | 33.1 (6.9) | 31.7 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 159 | 137 | 296
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 115 | 102 | 217
  Not Hispanic or Latino | 45 | 35 | 80
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 12 | 6 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 26 | 16 | 42
  White | 7 | 29 | 36
  More than one race | 4 | 5 | 9
  Unknown or Not Reported | 111 | 79 | 190
Region of Enrollment [Number; unit: participants]
  United States | 160 | 137 | 297
Nativity [Count of Participants; unit: Participants]
  US-born | 52 | 36 | 88
  Foreign-born | 108 | 101 | 209
Place of Birth (Foreign-Born) [Count of Participants; unit: Participants] — Population: Place of birth was assessed in the subgroup of participants who were foreign-born (n = 209).
  Participants
    number analyzed (Participants) | 108 | 101 | 209
    Dominican Republic | 57 | 12 | 69
    Ecuador | 2 | 25 | 27
    Mexico | 7 | 19 | 26
    Other birthplace | 42 | 45 | 87
Language Preference (Foreign-Born) [Count of Participants; unit: Participants] — Population: Language preference was assessed among the subgroup of participants who were foreign-born (n = 209).
  Participants
    number analyzed (Participants) | 108 | 101 | 209
    English | 24 | 22 | 46
    Spanish | 78 | 76 | 154
    Other | 6 | 3 | 9
Years in U.S. (Foreign-Born) [Mean (Standard Deviation); unit: years] — Population: Years in U.S. was assessed in the subgroup of participants who were foreign-born (n = 209).
  years
    number analyzed (Participants) | 108 | 101 | 209
    (all) | 10.4 (8.0) | 11.3 (7.3) | 10.9 (7.6)
Pregnancy Status [Count of Participants; unit: Participants]
  Not pregnant | 130 | 113 | 243
  Pregnant | 30 | 24 | 54
Breastfeeding Status [Count of Participants; unit: Participants]
  Not breastfeeding | 131 | 93 | 224
  Breastfeeding | 29 | 44 | 73
Educational Attainment [Count of Participants; unit: Participants]
  Some high school or less | 25 | 36 | 61
  High school diploma or equivalent | 57 | 46 | 103
  More than high school | 78 | 55 | 133
Car Ownership [Count of Participants; unit: Participants]
  Did not own a reliable car | 70 | 52 | 122
  Owned a reliable car | 90 | 85 | 175
Car Access: Ease of Borrowing a Car (If Not Owned) [Count of Participants; unit: Participants] — Population: Ease of borrowing a car was assessed among the subgroup of participants who did not own a car (n = 122).
  Participants
    number analyzed (Participants) | 70 | 52 | 122
    Very difficult | 41 | 14 | 55
    Difficult | 14 | 18 | 32
    Medium | 4 | 7 | 11
    Easy | 9 | 10 | 19
    Very Easy | 2 | 3 | 5
Car Access: How Often Can Use Car (If Owned) [Count of Participants; unit: Participants] — Population: How often can use car was assessed in the subgroup of participants who owned a car (n = 175).
  Participants
    number analyzed (Participants) | 90 | 85 | 175
    Never | 10 | 6 | 16
    Rarely | 3 | 6 | 9
    Sometimes | 14 | 12 | 26
    Often | 8 | 14 | 22
    Always | 55 | 47 | 102
Supplement Use [Count of Participants; unit: Participants]
  Not taking supplements | 84 | 61 | 145
  Taking supplements | 76 | 76 | 152
Smoking Status [Count of Participants; unit: Participants]
  Not at all | 147 | 127 | 274
  Some days | 7 | 2 | 9
  Every day | 3 | 4 | 7
  Not reported | 3 | 4 | 7
Past 7-Day Exposure to Secondhand Smoke [Count of Participants; unit: Participants]
  No | 127 | 124 | 251
  Yes | 33 | 11 | 44
  Not reported | 0 | 2 | 2
Food Security Status [Count of Participants; unit: Participants]
  Food secure | 91 | 83 | 174
  Food insecure | 65 | 53 | 118
  Not reported | 4 | 1 | 5
Meeting Physical Activity Guidelines [Count of Participants; unit: Participants]
  No | 59 | 64 | 123
  Yes | 101 | 73 | 174
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] — Height and weight were measured by trained research staff with participants wearing light clothing without shoes. Body mass index was calculated as weight in kilograms divided by height in square meters. Population: Because weight and height were measured at the time of study entry, among pregnant participants, weight and height before pregnancy, and correspondingly, pre-pregnancy BMI could not be determined. Pregnant women (n = 54) were therefore excluded from analyses of BMI (analysis sample size= 242).
  kg/m2
    number analyzed (Participants) | 129 | 113 | 242
    (all) | 29.5 (6.8) | 29.4 (6.8) | 29.4 (6.8)
Weight Status [Count of Participants; unit: Participants] — Based on their body mass index, participants were classified according to Centers for Disease Control and Prevention (CDC) weight status categories. Population: Because weight and height were measured at the time of study entry, among pregnant participants, weight and height before pregnancy, and correspondingly, pre-pregnancy BMI could not be determined. Pregnant women (n = 54) were therefore excluded from analyses of weight status (analysis sample size= 242).
  Participants
    number analyzed (Participants) | 129 | 113 | 242
    Underweight (BMI < 18.5) | 4 | 3 | 7
    Normal (BMI 18.5 to < 25) | 28 | 26 | 54
    Overweight (BMI 25 to < 30) | 44 | 44 | 88
    Obese (BMI ≥ 30) | 53 | 40 | 93
Social Desirability Trait [Mean (Standard Deviation); unit: units on a scale] — Assessed with a 5-item measure of socially desirable response set (SDRS-5). Response options are on a 5 point scale ranging from definitely true (1) to definitely false (5). Extreme SDRS responses are scored 1, and all other responses are scored 0. Responses are summed across items to derive a total score (score range 0-5). Higher scores indicate a worse outcome (the tendency to give socially desirable responses on self-report measures).
  units on a scale | 1.41 (1.75) | 3.22 (1.51) | 2.25 (1.88)
Children in the Household Aged 2-5 Years [Count of Participants; unit: Participants]
  None | 28 | 28 | 56
  One | 119 | 97 | 216
  Two | 13 | 12 | 25
Vegetable Intake Carotenoid Scores [Mean (Standard Deviation); unit: units on a scale] — Vegetable intake was objectively assessed using a reflection spectroscopy device (the Veggie Meter) to measure the level of carotenoid pigments in participants' skin (scores can range from 0 to 800). Higher scores indicate a better outcome (higher carotenoid levels).
  units on a scale | 265.17 (87.57) | 274.61 (105.5) | 269.54 (96.24)
Self-Reported Vegetable Intake [Mean (Standard Deviation); unit: Cups per day of vegetables consumed] | 1.46 (1.07) | 1.52 (1.07) | 1.49 (1.07)

OUTCOME MEASURES:

1. Primary Outcome: Vegetable Intake Carotenoid Scores at 3 Months
Description: Vegetable intake was objectively assessed using a reflection spectroscopy device (the Veggie Meter) to measure the level of carotenoid pigments in participants' skin (scores can range from 0 to 800). Higher scores indicate a better outcomes (higher carotenoid levels).
Time Frame: 3 months
Population: For vegetable intake carotenoid scores, analysis sample sizes were 137 in the intervention group and 124 in the control group. In the intervention group, 13 of the original 160 participants competed the baseline assessment only, 4 moved out of the area, and 6 discontinued their study involvement. In the control group, 10 of the original 137 participants completed the baseline assessment only, 2 moved out of the area, and 1 discontinued their study involvement).
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 137 | 124
units on a scale | 227.11 (9.91) | 269.98 (10.06)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.001, Mixed Models Analysis; Mean Difference (Net) = -42.87, 95% CI 2-sided [-65.25 to -20.49]

2. Primary Outcome: Vegetable Intake Carotenoid Scores at 6 Months
Description: as for outcome 1
Time Frame: 6 months
Population: For vegetable intake carotenoid scores, sample sizes were 137 in the intervention group and 124 in the control group. In the intervention group, 13 of the original 160 participants competed the baseline assessment only, 4 moved out of the area, and 6 discontinued their study involvement. In the control group, 10 of the original 137 participants completed the baseline assessment only, 2 moved out of the area, and 1 discontinued their study involvement.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 137 | 124
units on a scale | 236.01 (9.77) | 212.10 (9.79)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.031, Mixed Models Analysis; Median Difference (Net) = 23.91, 95% CI 2-sided [2.21 to 45.62]

3. Primary Outcome: Self-Reported Vegetable Intake at 3 Months
Description: Assessed with one of two items in a screening instrument developed by the National Cancer Institute. Participants reported the number of cups of vegetables (including 100% vegetable juice) they ate or drank each day (range 0-7). Higher numbers represent a better outcome (higher cups/day of vegetables consumed).
Time Frame: 3 months
Measure: Mean (Standard Error); unit: Cups per day
Arm/Group | Intervention | Control
Number analyzed (Participants) | 143 | 130
Cups per day | 1.78 (0.11) | 1.84 (0.12)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.662, Mixed Models Analysis; Median Difference (Net) = -0.06, 95% CI 2-sided [-0.33 to 0.21]

4. Primary Outcome: Self-Reported Vegetable Intake at 6 Months
Description: as for outcome 3
Time Frame: 6 months
Measure: Mean (Standard Error); unit: Cups per day
Arm/Group | Intervention | Control
Number analyzed (Participants) | 143 | 130
Cups per day | 1.83 (0.11) | 1.55 (0.12)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.047, Mixed Models Analysis; Mean Difference (Net) = 0.28, 95% CI 2-sided [0.00 to 0.55]

5. Primary Outcome: Number of Participants Who Redeemed Any Farmers' Market Nutrition Program (FMNP) Vouchers at 6 Months
Description: Objectively assessed using data provided by the collaborating WIC agency. WIC reported whether participants redeemed any FMNP vouchers (yes or no) from baseline to 6 months.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 160 | 137
Participants | 139 | 38
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p < 0.01, Regression, Logistic; Odds Ratio (OR) = 17.39, 95% CI 2-sided [8.64 to 35.02]

6. Secondary Outcome: Knowledge of Vegetable Intake Recommendations at 3 Months
Description: Assessed via self-report with an item from the National Cancer Institute's Food, Attitudes, and Behaviors (FAB) survey. Based on their responses, participants were classified as knowledgeable of the recommended cups per day (yes or no).
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 143 | 130
Participants | 10 | 4
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.056, Mixed Models Analysis; Odds Ratio (OR) = 3.9, 95% CI 2-sided [1.0 to 16.1]

7. Secondary Outcome: Knowledge of Vegetable Intake Recommendations at 6 Months
Description: as for outcome 6
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 143 | 130
Participants | 10 | 4
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.050, Mixed Models Analysis; Odds Ratio (OR) = 4.0, 95% CI 2-sided [1.0 to 16.3]

8. Secondary Outcome: Home Vegetable Availability (Quantity) at 3 Months
Description: Assessed with items from the Healthy Home Survey. Participants reported the number of fresh, frozen, and canned vegetables they had at home. Responses were summed across items to derive a total score (range 0-23). Higher scores indicate a better outcome (a higher number of vegetables at home).
Time Frame: 3 months
Measure: Mean (Standard Error); unit: Number of vegetables at home
Arm/Group | Intervention | Control
Number analyzed (Participants) | 143 | 130
Number of vegetables at home | 5.3 (0.3) | 7.1 (0.3)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.001, Mixed Models Analysis; Mean Difference (Net) = -1.7, 95% CI 2-sided [-2.5 to -1.0]

9. Secondary Outcome: Home Vegetable Availability (Quantity) at 6 Months
Description: as for outcome 8
Time Frame: 6 months
Measure: Mean (Standard Error); unit: Number of vegetables at home
Arm/Group | Intervention | Control
Number analyzed (Participants) | 143 | 130
Number of vegetables at home | 5.6 (0.3) | 6.3 (0.3)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.082, Mixed Models Analysis; Median Difference (Net) = -0.7, 95% CI 2-sided [-1.4 to 0.1]

10. Secondary Outcome: Home Vegetable Availability (Variety) at 3 Months
Description: Assessed with items from the Healthy Home Survey. Participants reported the number of fresh, frozen, and canned vegetables they had at home. The number of different (unique) vegetables reported was summed across items to derive a total score (range 0-21). Higher scores indicate a better outcome (a greater variety of vegetables at home).
Time Frame: 3 months
Measure: Mean (Standard Error); unit: Number of different vegetables at home
Arm/Group | Intervention | Control
Number analyzed (Participants) | 143 | 130
Number of different vegetables at home | 5.0 (0.3) | 6.5 (0.3)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.001, Mixed Models Analysis; Mean Difference (Net) = -1.5, 95% CI 2-sided [-2.2 to -0.8]

11. Secondary Outcome: Home Vegetable Availability (Variety) at 6 Months
Description: Assessed with items from the Healthy Home Survey. Participants reported the number of fresh, frozen, and canned vegetables they had at home. The number of different (unique) vegetables reported was summed to derive a total score (range 0-21). Higher scores indicate a better outcome (a greater variety of vegetables at home).
Time Frame: 6 months
Measure: Mean (Standard Error); unit: Number of different vegetables at home
Arm/Group | Intervention | Control
Number analyzed (Participants) | 143 | 130
Number of different vegetables at home | 5.2 (0.3) | 5.9 (0.3)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.039, Mixed Models Analysis; Median Difference (Net) = -0.7, 95% CI 2-sided [-1.4 to -0.0]

12. Secondary Outcome: Vegetable Taste Preferences at 3 Months
Description: Assessed with a single item (the Preference Rating Measure) querying overall, how much the participant likes the taste of vegetables (on a 7-point scale ranging from not at all to a lot). Scores can range from 1 to 7. Higher scores represent a better outcome (stronger vegetable taste preferences).
Time Frame: 3 months
Measure: Mean (Standard Error); unit: score on a 7-point scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 143 | 130
score on a 7-point scale | 6.3 (0.1) | 6.3 (0.1)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.962, Mixed Models Analysis; Mean Difference (Net) = -0.0, 95% CI 2-sided [-0.3 to 0.3]

13. Secondary Outcome: Vegetable Taste Preferences at 6 Months
Description: as for outcome 12
Time Frame: 6 months
Measure: Mean (Standard Error); unit: score on a 7-point scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 143 | 130
score on a 7-point scale | 6.3 (0.1) | 6.5 (0.1)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = .277, Mixed Models Analysis; Mean Difference (Net) = -0.2, 95% CI 2-sided [-0.4 to 0.1]

14. Secondary Outcome: Vegetable Preparation Practices at 3 Months
Description: Assessed via items from the Eating Among Teens and Young Adults Study (EAT)-II Survey (Laska et al., 2011). Participants reported how often, in the past month, they 1) bought fresh vegetables, 2) prepared a vegetable salad, and 3) prepared a dinner with vegetables. Responses were on a 5-point scale ranging from never to more than once a week. Ratings were summed across items to derive a total score. Scores can range from 1 to 15. Higher scores represent a better outcome (frequent use of the practices).
Time Frame: 3 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 143 | 130
units on a scale | 12.6 (0.2) | 13.0 (0.2)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.155, Mixed Models Analysis; Median Difference (Net) = -0.4, 95% CI 2-sided [-1.0 to 0.2]

15. Secondary Outcome: Vegetable Preparation Practices at 6 Months
Description: as for outcome 14
Time Frame: 6 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 143 | 130
units on a scale | 12.5 (0.2) | 12.4 (0.2)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.740, Mixed Models Analysis; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.5 to 0.7]

16. Secondary Outcome: Vegetable Preparation Skills at 3 Months
Description: Assessed via a single item (the Preparation Skills Rating Measure) querying how the participant would rate his or her overall skill in preparing vegetables (on a 7-point scale ranging from poor to excellent). Scores can range from 1 to 7. Higher scores represent a better outcome (greater vegetable preparation skills).
Time Frame: 3 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 143 | 130
units on a scale | 5.7 (0.1) | 6.0 (0.1)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = .122, Mixed Models Analysis; Median Difference (Net) = -0.2, 95% CI 2-sided [-0.5 to 0.1]

17. Secondary Outcome: Vegetable Preparation Skills at 6 Months
Description: as for outcome 16
Time Frame: 6 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 143 | 130
units on a scale | 5.6 (0.1) | 5.8 (0.1)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = .177, Mixed Models Analysis; Mean Difference (Net) = -0.2, 95% CI 2-sided [-0.5 to 0.1]

18. Secondary Outcome: Social Support for Vegetable Consumption at 3 Months
Description: Assessed via a single item (the Social Support Rating Measure) querying how much others support the participant to consume vegetables (on a 7-point scale ranging from not at all to a lot). Scores can range from 1 to 7. Higher scores represent a better outcome (greater social support for vegetable consumption).
Time Frame: 3 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 143 | 130
units on a scale | 5.9 (0.2) | 5.8 (0.2)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.514, Mixed Models Analysis; Median Difference (Net) = 0.1, 95% CI 2-sided [-0.3 to 0.5]

19. Secondary Outcome: Social Support for Vegetable Consumption at 6 Months
Description: as for outcome 18
Time Frame: 6 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 143 | 130
units on a scale | 6.0 (0.2) | 5.9 (0.2)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.335, Mixed Models Analysis; Median Difference (Net) = 0.2, 95% CI 2-sided [-0.2 to 0.6]

20. Secondary Outcome: Self-efficacy for Vegetable Consumption at 3 Months
Description: Assessed with a validated measure used to evaluate the Stellar Farmers' Market program (Dannefer et al., 2015). Participants rated how much they agreed or disagreed with statements designed to measure confidence in the ability to prepare and consume fresh produce. Item ratings are on a 4-point scale ranging from strongly disagree (1) to strongly agree (4). Ratings were summed across items to derive a total score. Scores can range from 5 to 20. Higher scores represent a better outcome (greater self-efficacy for vegetable consumption).
Time Frame: 3 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 143 | 130
units on a scale | 15.4 (0.2) | 15.3 (0.2)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.750, Mixed Models Analysis; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.4 to 0.6]

21. Secondary Outcome: Self-efficacy for Vegetable Consumption at 6 Months
Description: as for outcome 20
Time Frame: 6 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 143 | 130
units on a scale | 15.8 (0.2) | 16.0 (0.2)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.455, Mixed Models Analysis; Mean Difference (Net) = -0.2, 95% CI 2-sided [-0.7 to 0.3]

22. Secondary Outcome: Body Mass Index at 3 Months
Description: Height and weight were measured by trained research staff with participants wearing light clothing without shoes. Body mass index was calculated as weight in kilograms divided by height in square meters.
Time Frame: 3 months
Population: For weight status, sample sizes were 137 in the intervention group and 124 in the control group. In the intervention group, 13 of the original 160 participants competed the baseline assessment only, 4 moved out of the area, and 6 discontinued their study involvement. In the control group, 10 of the original 137 participants completed the baseline assessment only, 2 moved out of the area, and 1 discontinued their study involvement.
Measure: Mean (Standard Error); unit: kg/m2
Arm/Group | Intervention | Control
Number analyzed (Participants) | 137 | 124
kg/m2 | 30.3 (0.4) | 29.4 (0.4)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.053, Mixed Models Analysis; Mean Difference (Net) = 0.9, 95% CI 2-sided [-0.0 to 1.8]

23. Secondary Outcome: Body Mass Index at 6 Months
Description: as for outcome 22
Time Frame: 6 months
Population: as for outcome 22
Measure: Mean (Standard Error); unit: kg/m2
Arm/Group | Intervention | Control
Number analyzed (Participants) | 137 | 124
kg/m2 | 29.9 (0.4) | 29.9 (0.4)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = .986, Mixed Models Analysis; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.9 to 0.9]

24. Secondary Outcome: Number of Participants Who Met Physical Activity Guidelines at 3 Months
Description: Assessed with a validated 2-item measure (the Brief Physical Activity Assessment Tool or BPAAT [Marshall et al., 2005]). The instrument consists of two questions, one that assesses the frequency and duration of vigorous intensity physical activity and one that assesses the frequency and duration of moderate intensity physical activity undertaken in a usual week. A scoring algorithm is used to derive a total score (scores can range from 0 to 8). Participants are classified as meeting current physical activity guidelines (yes or no) based on the scores (a score greater than or equal to 4 indicates that the participant is meeting current physical activity guidelines, whereas a score between 0 and 3 indicates that the participant is not).
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 143 | 130
Participants | 94 | 83
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.810, Mixed Models Analysis; Odds Ratio (OR) = 1.1, 95% CI 2-sided [0.6 to 2.2]

25. Secondary Outcome: Number of Participants Who Met Physical Activity Guidelines at 6 Months
Description: Assessed with a validated 2-item measure (the Brief Physical Activity Assessment Tool or BPAAT [Marshall et al., 2005]). The instrument consists of two questions, one that assesses the frequency and duration of vigorous intensity physical activity and one that assesses the frequency and duration of moderate intensity physical activity undertaken in a usual week. A scoring algorithm is used to derive a total score (scores can range from 0 to 8). Participants are classified as meeting current physical activity guidelines (yes/no) based on the scores (a score greater than or equal to 4 indicates that the participant is meeting current physical activity guidelines, whereas a score between 0 and 3 indicates that the participant is not).
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 143 | 130
Participants | 97 | 91
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.591, Mixed Models Analysis; Odds Ratio (OR) = 0.8, 95% CI 2-sided [0.4 to 1.7]

26. Other Pre Specified Outcome: Number of Participants Who Redeemed Any Cash Value Vouchers or CVV at Farmers' Markets at 6 Months
Description: Objectively assessed using data provided by the collaborating WIC agency. WIC reported whether participants redeemed any cash value vouchers at farmers' markets (yes or no) between baseline and 6 months.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 160 | 137
Participants | 12 | 0

27. Other Pre Specified Outcome: Overall Satisfaction With Intervention
Description: Assessed via a single item (the Overall Satisfaction Rating Measure) querying how satisfied intervention recipients were with the intervention (on a 7-point scale ranging from very dissatisfied to very satisfied). Scores can range from 1 to 7. Higher scores represent a better outcome (greater overall satisfaction).
Time Frame: 6 months
Population: Satisfaction was measured among the subgroup of participants who received the intervention (n = 160). Of this number, 128 completed the measure of overall satisfaction with program.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 128 | 0
units on a scale | 6.8 (0.6) |

28. Other Pre Specified Outcome: Satisfaction With Intervention
Description: Assessed with a 5-item measure developed by the investigators querying how satisfied intervention recipients were with the intervention. Item responses were on a 7-point scale ranging from strongly disagree to strongly agree. Scores were averaged across items to derive a total score. Scores can range from 1 to7. Higher scores represent a better outcome (greater satisfaction with the intervention).
Time Frame: 6 months
Population: Satisfaction was measured among the subgroup of participants who received the intervention (n = 160). Of this number, 128 completed the satisfaction measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 128 | 0
units on a scale | 6.8 (0.5) |

ADVERSE EVENTS:
Time Frame: Adverse events were monitored over the course of participants' involvement in the study (the 34-week period beginning June 3, 2019, and ending January 31, 2020).
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/160 | 0/137
Serious Adverse Events (participants affected / at risk) | 0/160 | 0/137
Other Adverse Events (participants affected / at risk) | 0/160 | 0/137

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-19): https://cdn.clinicaltrials.gov/large-docs/85/NCT04038385/Prot_SAP_000.pdf